CLINICAL TRIAL: NCT03038477
Title: A Study of Durvalumab (MEDI4736), as an Adjuvant Therapy, Compared to Observation Alone, in Patients With Borderline Resectable Pancreatic Ductal Adenocarcinoma (BR PDA) Following Neoadjuvant Therapy and Successful Surgical Resection
Brief Title: A Study of Durvalumab in Patients With BR PDA Following Neoadjuvant Therapy and Successful Surgical Resection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cancelled by PI
Sponsor: University of Colorado, Denver (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0546.cc
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer
Keywords: Borderline Resectable Pancreatic Ductal Adenocarcinoma; Durvalumab
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Durvalumab (Experimental): Patients in Arm A will be given anti-PD-L1 antibody, durvalumab, every 2 weeks for a maximum of 26 doses if there is no radiographic evidence of disease recurrence. For Arm A, one cycle constitutes two durvalumab treatments on Day 1 and Day 15, respectively, repeated every 28 days.
  Interventions: Drug: Durvalumab
- No Durvalumab (No Intervention): Patients in Arm B will be observed.

INTERVENTIONS:
Drug: Durvalumab — 1500mg of Durvalumab will be given every 4 weeks (Q4W) for 12 months in patients enrolled in Arm A.
  Other Names: MEDI4736; anti-PD-L1 antibody
  Arms: Durvalumab

SUMMARY:
This is a two-arm, open-label, phase II study of in adult patients who have successfully undergone R0/R1 resection of PDAs following neoadjuvant chemotherapy and completion of adjuvant chemotherapy. Within 1-3 months of treatment completion, patients will be enrolled and randomized at a 1:1 ratio to receive durvalumab versus observation.

DETAILED DESCRIPTION:
Borderline resectable pancreatic cancer (BRPC) patients who have successfully underwent R0/R1 resection of PDAs following neoadjuvant chemotherapy, between 1-3 months after the completion of planned adjuvant chemotherapy will be enrolled and randomized at a 1:1 ratio into two arms (56 per arm). Patients in Arm A will be given anti-PD-L1 antibody, durvalumab, every 2 weeks for a maximum of 26 doses if there is no radiographic evidence of disease recurrence. Patients in Arm B will be observed. Blood draws for immune monitoring and serum banking will be collected at the following time points:

Arm A - before Cycles 1, 2, 4, 7 and End of Treatment (EOT) visit; Arm B - before Cycles 1, 4, 7, and End of Treatment (EOT) visit

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (e.g., HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age > 18 years at time of study entry, age > 20 years for Japanese subjects.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Life expectancy of > 2 years
5. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   * Absolute lymphocyte count ≥ 500/mm3
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). <<This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = (Weight (kg) x (140 - Age)) / (72 x serum creatinine (mg/dL))

   Females:

   Creatinine CL (mL/min) = (Weight (kg) x (140 - Age)) / (72 x serum creatinine (mg/dL)) x0.85
6. Women must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]).
7. Both women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must agree to use two (2) highly effective methods of contraception as outlined in this protocol for the duration of treatment with study drug plus 5 half-lives of study drug plus 90 days (duration of sperm turnover) for a total of 31 weeks post-treatment completion.
8. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
9. Have borderline resectable PDAs at the time of original diagnosis as per the AHPBA/SSO consensus on definition of borderline resectable PDA (see section 4.4 for definition of borderline resectable PDAs).
10. Have had an R0/R1 resection of PDA following neoadjuvant chemotherapy.
11. Have been more than one month and less than 3 months after the completion of planned adjuvant chemotherapy.
12. Have received at least one treatment of either FOLFIRINOX or gemcitabine/abraxane based regimens in both neoadjuvant and adjuvant setting. Neoadjuvant radiation is allowed.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrollment in the present study
2. Participation in another clinical study with an investigational product during the last 4 weeks.
3. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
4. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ
5. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 28 days prior to the first dose of study drug (≤ 28 days prior to the first dose of study drug for subjects who have received prior TKIs [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C). (If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period may be required.)
6. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
8. Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy).
9. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
10. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
11. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
12. History of primary immunodeficiency
13. History of allogeneic organ transplant
14. History of hypersensitivity to durvalumab or any excipient
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
16. Known history of previous clinical diagnosis of tuberculosis
17. History of leptomeningeal carcinomatosis
18. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
19. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
20. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
21. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
22. Subjects with uncontrolled seizures.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The number of subjects with disease free survival (DFS) | 26 Months
  Disease free survival (DFS) is defined as the time from randomization to the first of either disease recurrence or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) of all patients | 26 months
  OS is defined as the time from study enrollment to death from any cause.
The number of patients who experience adverse events | 26 months
  Adverse events are measured by Common Terminology Criteria for Adverse Events (CTCAE v4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No